CLINICAL TRIAL: NCT04558931
Title: An Open, Randomised, Controlled, Phase II Trial of CellProtect in Combination With Isatuximab Antibody Versus Isatuximab Antibody Alone as Maintenance Treatment in Patients With Multiple Myeloma Undergoing High Dose Treatment
Brief Title: Clinical Trial for Autologus NK Cells Alone or in Combination With Isatuximab as Maintenance for Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Sanofi (Industry); XNK Therapeutics AB, Sweden (Unknown)
Responsible Party: Principal Investigator, Hareth Nahi, M.D. PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISA-HC-NK
Record Dates: First submitted 2020-09-11; First posted 2020-09-22 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: NK cells; Consolidation; Isatuximab; SAR650984
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab

STUDY DESIGN:
Intervention Model Description: After confirmation of the eligibility criteria, patients will be randomly assigned in a 1:1 ratio to one of the two treatment arms:
  Isatuximab in combination with CellProtect (ISA/CellProtect experimental arm), or Isatuximab (ISA, control arm).
  Randomization will be at diagnosis and before the start of the treatment for patients eligible for SCT. Treatment administration will start within 100 days from AST date.
  Patients will be treated until disease progression (max 3 years), unacceptable adverse event (AE), patient's decision to stop the study treatment, death or any other reasons, whichever occurs first.
  Closing of randomization will occur after a total of approximately 60 patients have been randomized.
  After randomisation, patients in experimental arm will donate starting material for the production of the IMP.
  Manufacturing of CellProtect is promptly initiated for patients randomised to the active IMP arm A.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Isatuximab/CellProtect (Experimental): Isatuximab will be given intravenously (IV) at the dose of 10 mg/kg on Days 1, 8, 15, 22 (cycle 1), 36, 50 (cycle 2), 64, 78 (cycle 3) and monthly thereafter (cycles 4-36).
  CellProtect will be given IV infusion at the dose of 3x10^7 cells/kg day 29 , 43 and 3-10x10^7 on day 57.
  Each cycle will be 28 days, after completion of third cycles, patients will continue with Isatuximab alone until disease progression, unacceptable AE, death, completion of 3 years of treatment or patient's decision to discontinue, whichever occurs first.
  Interventions: Drug: CellProtect; Drug: Isatuximab
- B - Isatuximab (Active Comparator): Isatuximab will be given intravenously (IV) at the dose of 10 mg/kg on Days 1, 8, 15, 22 (cycle 1), 36, 50 (cycle 2), 64, 78 (cycle 3) and monthly thereafter (cycles 4-36).
  Each cycle will be 28 days, after completion of third cycles, patients will continue with Isatuximab alone until disease progression, unacceptable AE, death, completion of 3 years of treatment or patient's decision to discontinue, whichever occurs first.
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: CellProtect — In vitro expanded and activated autologous NK cells
  Other Names: Autologous NK cell
  Arms: A - Isatuximab/CellProtect
Drug: Isatuximab — Naked immunoglobulin (Ig) G1 monoclonal antibody (mAb) that selectively binds to the human cell surface antigen molecule classified as cluster of differentiation (CD) 38
  Other Names: Sarclisa

SUMMARY:
Prospective, single center, randomized, open label, parallel group, 2-arm study assessing the clinical benefit in term of enhancement of overall response rate of Isatuximab in combination with CellProtect as compared to Isatuximab for the treatment of patients with newly diagnosed multiple myeloma who are eligible for stem cell transplantation (SCT) as maintenance after SCT.

ELIGIBILITY:
Inclusion Criteria:

I1. Active multiple myeloma, as defined by the IMWG criteria.

I2. Evidence of measurable disease:

I3. Serum monoclonal (M)-protein ≥1.0 g/dL measured using serum protein immunoelectrophoresis a.and/or I4. Urine M-protein ≥200 mg/24 hours measured using urine protein immunoelectrophoresis

a. and/or I5. in patients without measurable M protein in serum or urine as per previous criteria, serum immunoglobulin free light chain (sFLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio <0.26 or >1.65.

I6. Patients who are newly diagnosed and considered for high-dose chemotherapy I7. Patient has given voluntary written informed consent before performance of any study related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to his/her medical care.

I8. ≥18 years of age (and satisfying the legal age of consent in the jurisdiction in which the study is taking place) I9. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 I10. Male or Female

1. Male participants A male participant must agree to use contraception of this protocol during the intervention period and for at least 5 months after the last dose of study treatment and refrain from donating sperm during this period.
2. Female participants

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

Not a Females of childbearing potential (FCBP), OR A FCBP who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting study medication and must either commit to continue abstinence from heterosexual intercourse or apply a highly effective method of birth control until at least 5 months after last dose of study treatment

Screening #2 (Conducted after HDT):

Inclusion criteria as for first screening in addition to response evaluation (at least partial remission must be met).

Exclusion Criteria:

E1. Prior or concurrent exposure to NK cells and NK like T cells, or Approved or investigational treatments for MM.

E2. Received any investigational drug within 14 days or 5 half-lives of the investigational drug, whichever is longer.

E3. Diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma (asymptomatic multiple myeloma with absence of related organ or tissue impairment end organ damage).

E4. Diagnosis of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.

E5. Prior or current systemic therapy, or SCT for symptomatic multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for 4 days) of corticosteroids, if completed within 14 days prior to randomization.

E6. Concomitant plasma cell leukemia. E7. Any major procedure within 14 days before the initiation of the study treatment: plasmapheresis, major surgery (kyphoplasty is not considered a major procedure), radiotherapy (except if palliative intent).

E8. ECOG PS >2. E9. Hemoglobin <8 g/dL. E10. Platelets <70 × 109/L if <50% of bone marrow (BM) nucleated cells are plasma cells, and ≤30 × 109/L if ≥50% of BM nucleated cells are plasma cells. Platelet transfusion is not allowed within 3 days before the screening haematological test.

E11. Total bilirubin >1.5 × upper limit of normal (ULN), except for known Gilbert syndrome.

E12. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3 × ULN.

E13. Hypersensitivity (or contraindication) to dexamethasone, sucrose histidine (as base and hydrochloride salt), boron, mannitol, and polysorbate 80 or any of the components of study therapy that are not amenable to premedication with steroids, pregelatinized starch, sodium stearyl fumarate, arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study therapy that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.

E14. Any of the following within 6 months prior to randomization:

E15. Second/third degree heart block E16. Poorly controlled hypertension E17. Myocardial infarction E18. Severe/unstable angina pectoris E19. Coronary/peripheral artery bypass graft E20. New York Heart Association class III or IV congestive heart failure E21. Grade ≥3 arrhythmias E22. Stroke or transient ischemic attack. E23. Left-ventricular ejection fraction <40%. E24. Prior malignancy. Adequately treated basal cell or squamous cell skin, or superficial (pTis, pTa, and pT1) bladder cancer, or low risk prostate cancer, or any in situ malignancy after curative therapy are allowed, as well as any other cancer for which cytotoxic chemotherapy has been completed ≥3 years prior to enrolment and from which the patient has been disease-free for ≥3 years.

E25. Known acquired immunodeficiency syndrome (AIDS)-related illness or known HIV disease requiring antiviral treatment or active hepatitis A (defined as positive HA antigen), B (defined as either positive HBs antigen or negative HBs antigen with positive HBc antibody), or C infection (defined as a known positive hepatitis C antibody result and known quantitative hepatitis C (HCV) ribonucleic acid (RNA) results greater than the lower limits of detection of the assay).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate as the occurrence of very good partial response or better after maintenance start | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 months
  Evaluate in both arms the occurance after maintenance start of: Very good partial response (VGPR) or better rate, as defined by the International Myeloma Working Group (IMWG) criteria.
Change in minimal residual disease (MRD) negativity rate | Before start of maintenance, after first Isatuximab cycle, before start of 4th Isatuximab cycle and at 12 and 24 months after start of maintenance
  Assessment of changes in MRD negativity rate in patients with complete and very good partial response as well as conversion of MRD positivity to MRD negativity.

SECONDARY OUTCOMES:
adverse events | From first dose of study treatment up to 30 days after the last dose of study treatment or initiation of further anti-myeloma therapy, whichever occurs first, assessed up to 96 months
  Assessment of treatment-emergent adverse events/serious adverse events (TEAEs/SAEs) (including IARs), laboratory parameters, vital signs, weight, ECOG PS, and findings from physical examination. TEAEs are defined as AEs that develop, worsen (according to the Investigator opinion), or become serious during the treatment period.
Time to progression | From date of first treatment until date of first documented progression, date of further anti-myeloma therapy or date of death from any cause, whichever came first, assessed up to 96 months
  The time from randomization to the date of first documentation of PD (as determined by the IRC using the IMWG criteria
Progression-free survival on/after study medication | From date of first treatment until date of first documented progression, date of further anti-myeloma therapy or date of death from any cause, whichever came first, assessed up to 96 months
  The time from the date of the start of maintenance treatment to the date of documented progressive disease (PD) or death, whichever comes first.
Duration of response | From date of first treatment until date of first documented progression, date of further anti-myeloma therapy or date of death from any cause, whichever came first, assessed up to 96 months
  The time from the date of the first IRC determined response to the date of first IRC PD or death, whichever occurs first. Duration of response will determined only for patients who have achieved CR, VGPR, or PR.
Overall survival | From date of first treatment until date of death from any cause, assessed up to 96 months
  Defined as the time from the date of randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Johan Lund, M.D., Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden